CLINICAL TRIAL: NCT03553290
Title: Lower-level Laser for Treating Dentinal Hypersensitivity
Brief Title: Therapeutic Evaluation of Lower-level Laser for Treating Dentinal Hypersensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 201701057DIPA
Record Dates: First submitted 2017-08-15; First posted 2018-06-12 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-03

CONDITIONS: Dentinal Hypersensitivity
Keywords: Dentistry; Dentinal Hypersensitivity; lower-level laser therapy

STUDY DESIGN:
Intervention Model Description: Split-mouth design in the same individual
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor were blinded from the arrangement of the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Sham Comparator): Mechanical debridement alone
  Interventions: Procedure: Control
- lower-level laser Therapy (Active Comparator): Mechanical debridement with lower-level laser therapy
  Device: A.R.C. FOX Laser-FOX Q-810nm Mechanical debridement with lower-level laser therapy
  Interventions: Device: A.R.C. FOX Laser-FOX Q-810nm

INTERVENTIONS:
Device: A.R.C. FOX Laser-FOX Q-810nm — 805-810 nm dichotomous laser, 12 Watt within the power of sensitive parts of the affected teeth
  Arms: lower-level laser Therapy
Procedure: Control — Mechanical debridement alone
  Arms: control

SUMMARY:
The aim of this study was to evaluate the efficacy of low energy laser for the treatment of dentinal hypersensitivity due to periodontal therapy.

DETAILED DESCRIPTION:
We will recruit 80 adult patients with obvious symptom of hypersensitivity after periodontal therapy. They will receive low-energy laser treatment, and the area without the symptom of hypersensitivity will be served as control. Changes in pain status and clinical periodontal index within six months of treatment will be recorded.

ELIGIBILITY:
Inclusion criteria

1.20-80 year-old with their own will and oral cleaning ability 2.Patients who have been diagnosed with periodontitis and have completed periodontal treatment 3.Gingival recession in at least two regions showed sensitivity of teeth (VAS> 5) 4.No systemic infection 5.No painkillers in the past two weeks 6.Not pregnant or lactating

Exclusion criteria

1.Smoking more than half a pack a day in the past month

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in mental status | 6 months
  Visual analogue scale analysis with a score range of 0-10 (0: no discomfort; 10: severe discomfort). Lower score represent a better outcome.

SECONDARY OUTCOMES:
Change in probing depth | 6 months
  Measure at six surfaces of tooth
Change in clinical attachment level | 6 months
  Measure at six surfaces of tooth
Change in gingival recession | 6 months
  Measure at six surfaces of tooth
Change in masticatory mucosa | 6 months
  Measure at mid-buccal aspect of tooth

CONTACTS AND LOCATIONS:
Overall Officials: Po-Chun Chang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan